## **HEALEY ALS Platform Trial - Regimen B Verdiperstat**

NCT04436510

**Document Date: 22 Jul 2022** 

### RGB REGIMEN-SPECIFIC STATISTICAL ANALYSIS PLAN (R-SAP)

**Master Protocol** Platform Trial for the Treatment of Amyotrophic Lateral

Sclerosis (ALS): A perpetual multi-center, multi-regimen,

clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS

**Regimen** RGB: Verdiperstat

Regimen Partner Biohaven Pharmaceuticals, Inc

**Regulatory Sponsor** Merit E. Cudkowicz, MD

**Master Protocol Version** 4.0, 31 Aug 2020

**RSA Version** 6.0, 02 Dec 2021

Master SAP Version 1.0, 24 Jun 2020

**R-SAP Version** 3.0, 22 Jul 2022

#### SAP APPROVAL SIGNATURES

DocuSigned by Merit Cudkowicz

| Merit Cudkowicz | I approve this document 07/22/2022 7:22:03 PM EDT | 07/22/2022 |
|---|---|---|
| Merit E. Cudkowicz M<br>Principal Investigator ar | Date | |
| —DocuSigned by Sabrina Pa | aganoni | |
| Sabrina Paganoni | 07/22/2022 | |
| Sabrina Paganoni: MD <sub>2</sub><br>Co-Principal Investigate | Date | |
| DocuSigned by Daniel Can | npbell | |
| Danul Campbell | 07/24/2022 | |
| Daniel Campbell PhD | 92BFDD76701C8<br>Biohaven Pharmaceuticals, Inc | Date |

DocuSigned by Ben Saville

Ben Saville

I approve this document 07/22/2022 | 6:27:55 PM EDT 07/22/2022

Beh-Saville PhD 432B98632C6FEC7283AD

Date

Senior Statistical Scientist, Berry Consultants

DocuSigned by Eric A. Macklin



Eric A. Macklin

| I approve this document | 07/22/2022 | 6:00:29 PM EDT

07/22/2022

Eric A Macklin 5 PhD 334DFC089673751 Study Biostatistician Date

## SAP REVISION HISTORY

| Version | Date | Description of Changes |
|---|---|---|
| 1.0 | 17 Mar 2022 | Initial version |
| 2.0 | 06 May 2022 | Revision of Section 5.9 Survival to specify that both PAV-free survival and overall survival will be evaluated at both the Week 24 Visit time point and the last-participant-last-visit time point and to specify that PAV-free survival to the Week 24 Visit time point is the primary analysis of survival in this analysis plan. |
| | | Revision of Section 6.5.5 CAFS to specify the following: |
| | | 1. CAFS will be used as a supportive analysis for the secondary efficacy endpoints of HHD upper and lower extremity percentage and SVC, |
| | | 2. Additional CAFS analyses will use multiple imputation to extend follow-up for participants who early terminate, withdraw consent, or are lost to follow-up, |
| | | 3. Additional CAFS analyses will use time to death alone independent of any death equivalent, and |
| | | 4. Primary inference from CAFS analyses will compare survival by time to death or death equivalent and will compare change in function to the last jointly observed time point. |
| 3.0 | 22 Jul 2022 | Revision of Section 4.2 Exploratory Endpoints to identify serum creatinine and serum and CSF neurofilament light chain (NfL) as exploratory biomarkers of neurodegeneration and neuromuscular degeneration and to include ALSAQ-40 domain scores and symptom index (SI) as exploratory endpoints. |
| | | Revision of Section 5.1 ALSFRS-R to specify details of the calculation of pre-baseline slope. |
| | | Revision of Section 5.5 Quantitative Voice Characteristics to include predicted vital capacity as an additional metric at the Baseline Visit. |
| | | Revision of Section 5.6 Biofluid Biomarkers of Neurodegeneration to specify the assay techniques used to quantify serum creatinine and serum and CSF NfL and to specify that levels of serum and CSF NfL will be log-transformed in all analyses. |

| Version | Date | Description of Changes |
|---|---|---|
| 3.0 (continued) | 22 Jul 2022<br>(continued) | Revision of Section 5.7 ALSAQ-40 to specify calculation of domain scores and to revise calculation of overall ALSAQ-40 SI. |
| | | Revision of Section 5.8 CNS-BFS to specify that the total score is referenced. Revision of Section 5.9 Survival to specify that time at risk begins at each participant's Baseline Visit and to specify that the date of PAV initiation, where applicable, will be imputed as the fifteenth day of a month if not specified more precisely. |
| | | Revision of Section 6.1 Analysis Sets to add the Efficacy Common Mode of Administration (ECM) analysis set, to remove the restriction on protocol deviations that could be considered for exclusion from the Efficacy Per-protocol (EPP) analysis set must be classified as major protocol deviations, to specify the time point at which data is excluded from the EPP analysis set in the case of time-dependent exclusions, and to specify that data from placebo participants from other regimens would not be excluded from the EPP analysis set due to non-adherence to protocol-specified dosing. |
| | | Revision of Section 6.2 Baseline Characterization to include ALSAQ-40 domain scores and SI. |
| | | Revision of Section 6.5.2 Repeated-measures Model to add a fixed term for treatment group (removing the shared-baseline assumption at the recommendation of the FDA) and to specify a separate supportive analysis that includes fixed terms for centered baseline serum NfL level and centered baseline serum NfL level × visit interaction. |
| | | Revision of Section 6.5.3 Random-slopes Model to add a fixed term for treatment group (removing the shared-baseline assumption) and to specify a separate supportive analysis that includes fixed terms for centered baseline serum NfL level and centered baseline serum NfL level × study month interaction. |
| | | Revision of Section 6.5.4 Survival and Time to Clinical Events to clarify that survival analyses that include follow-up beyond the placebo-controlled period will be analyzed in the ERO analysis set, to include baseline age as an additional covariate in all adjusted models, and to specify an additional adjusted analysis that includes baseline serum NfL level as a covariate. |

| Version | Date | Description of Changes |
|---|---|---|
| 3.0 (continued) | 22 Jul 2022<br>(continued) | Revision of Section 6.5.5 CAFS to clarify that the primary CAFS analysis is specified in the ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report and to add two additional sets of CAFS analyses that adjust rank scores in linear models, one set that adjusts for time from ALS symptom onset, delta-FRS, baseline use of riluzole, and baseline use of edaravone, and one set that adjusts for the same set of covariates plus baseline serum NfL level. |
| | | Revision of Section 6.5.6 HHD0 and HHD0 <sup>2</sup> to remove reference to the shared-baseline assumption of the repeated-measures mixed model of Section 6.5.2 and to specify a separate analysis that adds baseline serum NfL level as an additional covariate. |
| | | Revision of Section 6.5.7 Quantitative Voice Measures to remove reference to the shared-baseline assumption of the random-slopes mixed model of Section 6.5.3 and to add a fixed term for treatment group (removing the shared-baseline assumption) and to specify a separate analysis that includes fixed terms for centered baseline serum NfL level and centered baseline serum NfL level × B-spline interaction. |
| | | Revision of Section 6.5.8 Placebo Multiple Imputation to specify regression over sequential visits by the fully conditional specification method, to remove reference to the shared-baseline assumption of the repeated-measures mixed model of Section 6.5.2, and to specify a separate analysis that adds baseline serum NfL level as an additional covariate. |
| | | Revision of Section 6.5.11 Comparison of Controls across<br>Regimens to specify separate analyses that add baseline serum<br>NfL level as an additional covariate. |

#### **ABBREVIATIONS**

ALP Alkaline Phosphatase

ALS Amyotrophic Lateral Sclerosis

ALSAQ-40 Amyotrophic Lateral Sclerosis Assessment Questionnaire, 40-item version

ALSFRS-R Amyotrophic Lateral Sclerosis Functional Rating Scale, Revised

ALT Alanine Transaminase
AST Aspartate Transaminase

ATC WHODrug Anatomical, Therapeutic, and Chemical class

ATS American Thoracic Society

BLQ Below the Limit of Quantitation

BMI Body Mass Index

C-SSRS Columbia Suicide Severity Rating Scale

CAFS Combined Assessment of Function and Survival

CBC Complete Blood Count
CKD Chronic Kidney Disease
COVID-19 Coronavirus Disease 2019

CNS-BFS Center for Neurologic Study Bulbar Function Scale

CSF Cerebrospinal Fluid
CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

delta-FRS Pre-baseline Slope in ALSFRS-R

DAP Data Analysis Plan

DILI Drug-induced Liver Injury
DNA Deoxyribonucleic Acid

DRR Disease Rate Ratio

ECC Efficacy Concurrent Control

ECG Electrocardiography or Electrocardiogram

eGFR Estimated Glomerular Filtration Rate

EPP Efficacy Per-protocol
ERO Efficacy Regimen-only

ELISA Enzyme-linked Immunosorbent Assay

FAS Full Analysis Set

### ABBREVIATIONS (continued)

FVC Forced Vital Capacity
GLI Global Lung Initiative

hCG Human Chorionic Gonadotropin

HHD Hand-held Dynamometry

HLT MedDRA High Level Term

ICF Informed Consent Form

ITT Intention-to-treat Principle

M-SAP Master Statistical Analysis Plan

MDRD Modification of Diet in Renal Disease

MedDRA Medical Dictionary for Regulatory Activities

MP Master Protocol

MPRDR ALS Master Protocol Recommended Statistical Analysis, Design and

Simulation Report

NCI National Cancer Institute

NEALS Northeast ALS

NfL Neurofilament Light Chain

NIV Noninvasive Ventilation

OLE Open-label Extension

PAV Permanent Assisted Ventilation

PD Pharmacodynamics

PK Pharmacokinetics

PT MedDRA Preferred Term

RBC Red Blood Cell

RDW RBC Distribution Width

RGB Regimen B (verdiperstat)

RSA Regimen-specific Appendix

R-SAP Regimen-specific Statistical Analysis Plan

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SGOT Serum Glutamic Oxaloacetic Transaminase

SGPT Serum Glutamic Pyruvic Transaminase

## ABBREVIATIONS (continued)

SI Symptom Index

SoA Schedule of Activities

SOC MedDRA System Organ Class

SRO Safety Regimen-only

STF Safety and Tolerability Full

STN Safety and Tolerability Narrow

SVC Slow Vital Capacity

TBL Total Bilirubin

TEAE Treatment-emergent Adverse Event

TSH Thyroid Stimulating Hormone

ULN Upper Limit of Normal

WBC White Blood Cell

WHODrug World Health Organization Drug Dictionary Enhanced

## **Table of Contents**

| 1. | | | ng Documents | |
|---|---|---|---|---|
| 2. | St | tudy Do | esign | 11 |
| | 2.1 | Overvi | ew | 11 |
| | 2.2 | Study ( | Objectives | 12 |
| | 2.3 | | Population | |
| | 2.4 | | pant Flow | |
| | 2.5 | | en Allocation | |
| | 2.6 | | ent Allocation | |
| | 2.7 | | ent Administration | |
| | 2.8 | | tion Concealment | |
| | 2.9 | | chedule of Activities (SoA) | |
| 3. | | | Considerations for Data Analysis | |
| ٠. | 3.1 | | cal Software | |
| | 3.2 | | ary Statistics | |
| | 3.3 | | on | |
| | 3.4 | | ormations | |
| | 3.5 | | licity Adjustments | |
| | 3.6 | | g Data | |
| 1 | | | | |
| 4. | | | idpoints | |
| | 4.1 | | y Endpoints | |
| | 4.2 | | atory Endpoints | |
| _ | 4.3 | | Endpoints | |
| 5. | | | ment Definitions | |
| | 5.1 | | S-R | |
| | 5.2 | | | |
| | 5.3 | | Spirometry | |
| | 5.4 | HHD a | nd Grip Strength | 17 |
| | 5.5 | | tative Voice Characteristics | |
| | 5.6 | Bioflui | d Biomarkers of Neurodegeneration | 18 |
| | 5.7 | ALSA | Q-40 | 18 |
| | 5.8 | CNS-B | FS | 18 |
| | 5.9 | Surviva | al | 18 |
| | 5.10 | Kin | g's ALS Clinical Staging System | 19 |
| | 5.11 | | pitalization and Other Clinical Events | |
| | 5.12 | | rmacodynamic Biomarkers | |
| | 5.13 | | ical Safety Laboratory Tests | |
| 6. | St | | al Methodology | |
| | 6.1 | | is Sets | |
| | - | | e Characterization | 22 |
| | 6.3 | Primar | y Efficacy Analysis and Supportive Analyses | 22 |
| | 6.4 | | Analysis | |
| | 6.5 | | lary Efficacy Analyses | |
| | | | Hierarchical Testing | |
| | | | Repeated-measures Model | |
| | | | Random-slopes Model | |
| | | | Survival and Time to Clinical Events | |
| | | | CAFS | |
| | | | HD0 and HHD0 <sup>2</sup> | |
| | | | Quantitative Voice Measures | |
| | | | Placebo Multiple Imputation. | |
| | | | Additional Sensitivity Analyses of Primary and Key Secondary Outcomes | |
| | | | Subgroup Analyses | |
| | | | Comparison of Controls across Regimens | |
| | 6 | 5.12 F | harmacokinetic Analyses | 30 |

| | 6.5.13 | Pharmacodynamic Biomarker Analyses | 30 |
|----|----------|------------------------------------------|----|
| | 6.6 Safe | ty Analyses | |
| | 6.6.1 | Treatment-emergent Adverse Events | |
| | 6.6.2 | Safety Labs | 31 |
| | 6.6.3 | ECG Results. | |
| | 6.6.4 | Vital Signs and Weight | 31 |
| | 6.6.5 | Suicidality | 31 |
| | 6.7 Othe | er Analyses | 32 |
| | 6.7.1 | Participant Disposition | 32 |
| | 6.7.2 | Study Drug Compliance and Tolerance | 32 |
| | 6.7.3 | Concomitant Medication Use | 33 |
| | 6.7.4 | Medical History | 33 |
| | 6.7.5 | Blindedness | 33 |
| | 6.7.6 | Protocol Deviations | 33 |
| | 6.7.7 | Impact of COVID-19 Pandemic | 33 |
| 7. | Valida | tion | |
| | 7.1 Prim | nary Efficacy Analysis | 33 |
| | | ondary, Exploratory, and Safety Analyses | |
| 8. | | ences | |

### 1. Governing Documents

This Regimen-specific Statistical Analysis Plan (R-SAP) for the verdiperstat regimen (RGB) specifies any modification from the default outcome measures, analysis samples, and planned analyses for the placebo-controlled period of the HEALEY ALS Platform Trial as specified in the Master SAP (M-SAP). The M-SAP and this R-SAP supplement the Master Protocol, the "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (Appendix 1 to the Master Protocol), and the RGB Regimen-specific Appendix (RSA). Please refer to the Master Protocol and the RGB RSA for details on the rationale for the study design, eligibility criteria, conduct of the trial, clinical assessments and schedule of assessments, definitions and reporting of adverse events, data management conventions, and regulatory oversight and compliance procedures. The "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (MPRDR) and any regimen-specific deviations described in the RGB RSA and this R-SAP are authoritative in defining the primary and interim analyses. In case of discrepancies between the RGB RSA and this R-SAP concerning use of shared placebos, this R-SAP is authoritative. In case of discrepancies between either SAP and the Master Protocol and the RGB RSA concerning matters of analysis other than the primary and interim analyses and use of shared placebos, the M-SAP and this R-SAP are authoritative. In case of discrepancies between the M-SAP and this R-SAP, this R-SAP is authoritative. On all matters not related to analysis, the Master Protocol and the RGB RSA are authoritative. The following table describes relationships among the relevant documents in adjudicating possible discrepancies with higher numbers indicating greater authority.

| Issues potentially requiring adjudication | Master<br>Protocol | RGB<br>RSA | MPRDR | M-SAP | RGB<br>R-SAP |
|---|---|---|---|---|---|
| Use of shared placebos | 1 | 4 | 2 | 3 | 5 |
| Primary and interim analysis specifications not related to use of shared placebo | 1 | 5 | 4 | 2 | 3 |
| Statistical analysis specifications not related to use of shared placebo or primary and interim analyses | 1 | 3 | 2 | 4 | 5 |
| All matters not related to statistical analysis | 4 | 5 | 1 | 2 | 3 |

### 2. Study Design

#### 2.1 Overview

The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. RGB evaluates the safety and efficacy of verdiperstat administered orally at a dosage of 600 mg BID vs. placebo. The RGB RSA describes the nature of the intervention and its mechanism of action, the mode and frequency of administration, additional eligibility criteria beyond those specified in the Master Protocol, additional enrollment procedures, and additions and modifications of safety and efficacy assessments relative to those outlined in the Master Protocol.


### 2.2 Study Objectives

Primary Efficacy Objective:

• To evaluate the efficacy of verdiperstat as compared to placebo on ALS disease progression.

Secondary Efficacy Objectives:

• To evaluate the effect of verdiperstat on selected secondary measures of disease progression, including survival.

Safety Objectives:

• To evaluate the safety of verdiperstat for ALS patients.

**Exploratory Efficacy Objectives:** 

- To evaluate the effect of verdiperstat on selected biomarkers and endpoints.
- To explore verdiperstat pharmacokinetics (PK) and pharmacodynamic (PD) effects.

## 2.3 Study Population

In addition to eligibility criteria specified in the Master Protocol, participants in RGB must not be taking strong inhibitors of CYP1A2 (i.e., ciprofloxacin, enoxacin, fluvoxamine, zafirlukast) or CYP3A4 (i.e., conivaptan, itraconazole, ketoconazole, posaconazole, troleandomycin, voriconazole, clarithromycin, diltiazem, idelalisib, nefazodone, and certain antiviral agents [cobicistat, danoprevir, ritonavir, elvitegravir, indinavir, lopinavir, paritaprevir, ombitasavir, dasabuvir, saquinavir, tipranavir, nelfinavir]) for chronic/long-term use, defined as more than two weeks.

Participants will be recruited from approximately 60 centers located throughout the US that are part of the Northeast ALS (NEALS) Consortium.

#### 2.4 Participant Flow

Participants in RGB follow the consenting, Master screening, regimen assignment, regimen-specific screening, randomization to active or placebo treatment, and follow-up procedures and timing described in the M-SAP. Detailed descriptions of study procedures and timing are specified in the Master Protocol and the RGB RSA.

#### 2.5 Regimen Allocation

Participants in RGB are those determined eligible for Master Protocol-level inclusion and exclusion criteria and randomly assigned to RGB, stratified by use of riluzole, edaravone, both, or neither at the time of screening for the Master Protocol. Details of regimen assignment are described in the Platform Trial Regimen Assignment Plan.

#### 2.6 Treatment Allocation

Participants in RGB are randomly allocated in a 3:1 ratio to active or placebo treatment based on a pre-specified permuted-block randomization schedule, stratified by use of riluzole, edaravone, both, or neither at the time of screening for the Master Protocol.

#### 2.7 Treatment Administration

Verdiperstat and placebo are supplied as matching reddish-beige, film coated, oval tablets. Each tablet of active study drug contains 300 mg of verdiperstat as the free base plus excipients generally recognized as safe for oral administration in an extended-release formulation.

The first dose of study drug should be administered while in the office/clinic on the day of the Baseline Visit after all visit assessments are complete. Participants should stay at the office/clinic for monitoring for approximately 30 minutes post-dose. From the Baseline Visit to the end of Week 1, participants should take one tablet of study drug per day. During Week 2, participants should take one tablet of study drug twice per day. Starting at the beginning of Week 3 and throughout the remainder of the study, participants should take two tablets of study drug twice per day. If tolerability issues are experienced, the titration schedule may be modified. If a participant is off study drug for more than 14 consecutive days, the participant should re-escalate using the titration paradigm described above.

Additional details of treatment administration are described in the RGB RSA.

### 2.8 Allocation Concealment

Allocation concealment is the same as described in the M-SAP.

### 2.9 RGB Schedule of Activities (SoA)

| | MP | RGB | Base- | Week | Week | | Week | Week | Week | | Final |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scrn <sup>1</sup> | Scrn <sup>1</sup> | line | <b>2</b> <sup>2</sup> | 4 <sup>18,19</sup> | 818,19 | 12 | 1618,19 | 20 | <b>24</b> <sup>3,18</sup> | Call <sup>3,4</sup> |
| | Cln | Cln | Cln | Phn | Cln <sup>5</sup> | Cln <sup>5</sup> | Phn | Cln <sup>5</sup> | Phn | Cln | Phn |
| | -42d | -41d | Day | Day | Day | Day | Day | Day | Day | Day | 28d ±3 |
| Activity | to -1d | to 0d | 0 | 14±3 | 28±7 | 56±7 | 84±3 | 112±7 | 140±3 | 168±7 | ALD |
| Written Informed Consent <sup>5</sup> | X | X | | | | | | | | | |
| Inclusion/Exclusion Review | X | $X^6$ | | | | | | | | | |
| ALS & Medical History | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Physical Examination | X | | | | | | | | | | |
| Neurological Exam | X | | | | | | | | | | |
| Vital Signs <sup>7</sup> | X | | X | | X | X | | X | | X | |
| Slow Vital Capacity | $X^{20}$ | | X | | | C | | С | | X | |
| Home Spirometry | $X^{20}$ | | X | | | X | | X | | X | |
| Muscle Strength Assessment | | | X | | | С | | C | | X | |
| ALSFRS-R | X | | X | | X | X | X | X | X | X | |
| ALSAQ-40 | | | X | | | | | | | X | |
| CNS-BFS | | | X | | | X | | X | | X | |
| 12-Lead ECG | X | | | | | С | | | | X | |
| Clinical Safety Labs <sup>8</sup> | X | | X | | X | X | | X | | X | |
| Verdiperstat PK Samples <sup>10</sup> | | | X | | C | C | | C | | X | |
| Verdiperstat PD Samples <sup>10</sup> | | | X | | C | С | | C | | X | |
| Biomarker Blood Collection | | | X | | | С | | С | | X | |
| Biomarker Urine Collection | | | X | | | C | | C | | X | |
| DNA Collection <sup>11</sup> (optional) | | | X | | | | | | | | |
| CSF Collection (optional) | | | X | | | | | C <sup>17</sup> | | | |
| Concomitant Medication Review | X | X | X | X | X | X | X | X | X | X | |
| Adverse Event Review <sup>9</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Suicidality C-SSRS | | | X | | X | X | | X | | X | |
| Install Smartphone Apps <sup>21</sup> | | | X | | | | | | | | |


| | MP | RGB | Base- | Week | Week | Week | Week | Week | Week | Week | Final |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scrn <sup>1</sup> | Scrn <sup>1</sup> | line | <b>2</b> <sup>2</sup> | 4 <sup>18,19</sup> | 818,19 | 12 | 1618,19 | 20 | 243,18 | Call <sup>3,4</sup> |
| | Cln | Cln | Cln | Phn | Cln <sup>5</sup> | Cln <sup>5</sup> | Phn | Cln <sup>5</sup> | Phn | Cln | Phn |
| | -42d | -41d | Day | Day | Day | Day | Day | Day | Day | Day | 28d ±3 |
| Activity | to -1d | to 0d | 0 | 14±3 | 28±7 | 56±7 | 84±3 | 112±7 | 140±3 | 168±7 | ALD |
| Smartphone Voice Recording <sup>12</sup> | | | X | | X | X | | X | | X | |
| Uninstall Smartphone App | | | | | | | | | | X | |
| Regimen Assignment | X | | | | | | | | | | |
| Randomization within RGB | | | X | | | | | | | | |
| Administer/Dispense Study Drug | | | $X^{13}$ | | X | X | | X | | | |
| Drug Accountability/Compliance | | | | $X^{2,22}$ | X | X | $X^{22}$ | X | $X^{22}$ | X | |
| Dose Escalation | | | $X^{15}$ | $X^{15}$ | | | | | | | |
| Exit Questionnaire | | | | | | | | | | X | |
| Vital Status | | | | | | | | | | $X^{16}$ | |

Abbreviations: ALD = after last dose, ALS = amyotrophic lateral sclerosis, ALSAQ-40 = ALS Assessment Questionnaire, ALSFRS-R = ALS Functional Rating Scale Revised, BP = blood pressure, C = completed only if the visit is conducted in-clinic, CBC = complete blood count, Cln = Clinic visit, CNS-BFS = Center for Neurologic Study Bulbar Function Scale, CSF = cerebrospinal fluid, C-SSRS = Columbia-Suicide Severity Rating Scale, d = day, DNA = deoxyribonucleic acid, ECG = electrocardiogram, LFTs = liver function tests, MP = Master Protocol, PD = pharmacodynamic, Phn = Phone visit, RGB = the verdiperstat regimen, Scrn = Screening Visit.

<sup>&</sup>lt;sup>1</sup> Master Protocol Screening procedures must be completed within 42 days to 1 day prior to the Baseline Visit. The Regimen-Specific Screening Visit and Baseline Visit should be combined if possible.

<sup>&</sup>lt;sup>2</sup> At the end of Week 2, an assessment of compliance and tolerance to this dose titration schedule will be conducted. The assessment will be conducted by phone. If tolerability issues are experienced with 300 mg QD or 300 mg BID dosing, the titration schedule may be modified (see RSA Section 5.3.2).

<sup>&</sup>lt;sup>3</sup> Participants will only have a Follow-Up Safety Call at this time if they do not continue into the OLE or if they discontinue prior to Week 24. Participants who continue into OLE will have a Follow-Up Safety Call after their last dose of study drug during the OLE phase.

<sup>&</sup>lt;sup>4</sup> Participants who continue into the OLE and then early terminate will be asked to complete an Early Termination Visit and Follow-Up Safety Call as described in the body of this RSA.

<sup>&</sup>lt;sup>5</sup> During the Master Protocol Screening Visit, participants will be consented via the Master Protocol informed consent form (ICF). After a participant is randomized to a regimen, participants will be consented a second time via the RSA ICF.

<sup>&</sup>lt;sup>6</sup> At the Regimen Specific Screening Visit, participants will have regimen-specific inclusion and exclusion criteria assessed, if applicable.

<sup>&</sup>lt;sup>7</sup> Vital signs include weight, systolic and diastolic pressure, respiratory rate, heart rate and temperature. Height is measured at Master Protocol Screening Visit only.

<sup>&</sup>lt;sup>8</sup> Clinical safety labs include hematology (CBC with differential), complete chemistry panel, thyroid function (TSH) and urinalysis. Serum pregnancy testing will occur in women of child-bearing potential at the Master Protocol Screening Visit and as necessary during the study. Pregnancy testing is only repeated as applicable if there is a concern for pregnancy.

<sup>&</sup>lt;sup>9</sup> Adverse events that occur after signing the master protocol consent form will be recorded.

<sup>&</sup>lt;sup>10</sup> Myeloperoxidase protein and activity, and plasma concentrations of verdiperstat will be measured. For each sample, the time of the last verdiperstat or matching placebo dose prior to sample collection, time of the last meal prior to sampling and time of the PD/PK sample collection should be reported on the CRF.

<sup>&</sup>lt;sup>11</sup> The DNA sample can be collected after baseline if a baseline sample is not obtained or the sample is not usable.

<sup>&</sup>lt;sup>12</sup> In addition to study visits outlined in the SOA, participants may be asked to complete twice weekly voice recordings at home. During weeks when a participant is doing a voice recording in-clinic, he or she would only do one other voice recording at home that week.

- <sup>16</sup> Vital status, defined as a determination of date of death or death equivalent or date last known alive, will be determined for each randomized participant at the end of the placebo-controlled portion of their follow-up (generally the Week 24 Visit, as indicated). If at that time the participant is alive, his or her vital status should be determined again at the time of the last participant's last visit of the placebo-controlled portion of a given regimen. We may also ascertain vital status at later time points by using publicly available data sources as described in section 8.15 of the Master Protocol.
- <sup>17</sup> If the CSF collection cannot happen at the Week 16 Visit for logistical reasons such as scheduling, it can happen at the Week 24 Visit.
- <sup>18</sup> Participants should be instructed to skip the morning dose of study drug on the day of the study visit. Study drug should not be taken until after study visit procedures are complete.
- <sup>19</sup> Visit may be conducted via phone or telemedicine with remote services instead of in-person if this is needed to protect the safety of the participant due to a pandemic or other reason.
- <sup>20</sup> If required due to pandemic-related restrictions, Forced Vital Capacity (FVC) performed by a Pulmonary Function Laboratory evaluator or with a study-approved home spirometer, or sustained phonation using a study approved method may be used for eligibility (Master Protocol Screening ONLY).
- <sup>21</sup> Two smartphone apps should be installed on the participant's phone, one to collect the voice recordings and one to collect home spirometry.
- <sup>22</sup> Drug accountability will not be done at phone visits. A drug compliance check in must be held during phone visits to ensure participant is taking drug per dose regimen and to note any report of missed doses.

### 3. General Considerations for Data Analysis

#### 3.1 Statistical Software

Statistical software use for analyses is the same as described in the M-SAP.

### 3.2 Summary Statistics

Data summaries are the same as described in the M-SAP.

#### 3.3 Precision

Precision of reported results is the same as described in the M-SAP.

#### 3.4 Transformations

Data transformations are the same as described in the M-SAP.

### 3.5 Multiplicity Adjustments

Handling of multiplicity adjustments is the same as described in the M-SAP.

<sup>&</sup>lt;sup>13</sup> Administer first dose of investigational product (IP) only after Baseline Visit procedures are completed. Participants should take the first dose of IP while in the office/clinic on the day of the Baseline visit and stay at the clinic for approximately 30 minutes post-dose for observation.

<sup>&</sup>lt;sup>14</sup> Investigational product will only be dispensed at this visit if the participant continues in the OLE.

<sup>&</sup>lt;sup>15</sup> From start to end of Week 1, participants will ingest either 300 mg QD of verdiperstat or matching placebo QD. From start to end of Week 2, participants will ingest either 300 mg BID of verdiperstat or matching placebo BID. Starting with Week 3 and continuing to Week 24, participants will ingest either 600 mg BID of verdiperstat or matching placebo BID.

### 3.6 Missing Data

Handling of missing data is the same as described in the M-SAP. Clinic-based assessments that are missing due to COVID-19 restrictions or disruptions are considered missing at random.

### 4. Study Endpoints

### 4.1 Efficacy Endpoints

The primary and secondary efficacy endpoints are the same as described in the M-SAP. ALSFRS-R total score is considered the primary efficacy endpoint and hand-held dynamometry (HHD) upper and lower extremity percentages, slow vital capacity (SVC), and survival are considered key secondary efficacy endpoints in RGB.

### 4.2 Exploratory Endpoints

The following categories of exploratory endpoints will be evaluated:

- Change in ALSFRS-R domain scores
- Change in strength: HHD global percentage, HHD0, and HHD0<sup>2</sup>,
- Change in quantitative voice characteristics as measured by Aural Analytics: maximum phonation time, pause rate, breathy vocal quality, pitch instability, regulation of voicing, articulatory precision, speaking rate, articulation rate, and monotonicity,
- Change in biofluid biomarkers of neurodegeneration and neuromuscular degeneration: serum creatinine and serum and cerebrospinal fluid (CSF) neurofilament light chain (NfL),
- Change in patient-reported outcomes: ALSAQ-40 physical mobility, independence in activities of daily living, eating and drinking, communications, and emotional reactions domain scores and ALSAQ-40 symptom index, CNS-BFS total score,
- Change in plasma concentrations of verdiperstat,
- Change in verdiperstat PD biomarkers: myeloperoxidase protein, total activity, and concentration-specific activity,
- Change in respiratory function as assessed by home spirometry, and
- Time to clinical events: first hospitalization due to a serious adverse event (SAE), first hospitalization due to an ALS-related SAE, first use of assisted ventilation, first placement of a feeding tube, first time reaching King's stage 4a or 4b, and first instance of any of the following events: hospitalization for an SAE, feeding tube placement, tracheostomy, initiation of permanent assisted ventilation (PAV), or death.

### 4.3 Safety Endpoints

In addition to the safety endpoints described in the M-SAP, the following RGB regimen-specific safety endpoint will be evaluated:

• Thyroid function: Proportion of participants with TSH ≥10 mIU/L, proportion of participants with signs or symptoms of hypothyroidism, and levels of free T3, free T4, and TSH.

#### 5. Measurement Definitions

#### 5.1 ALSFRS-R

The definitions of ALSFRS-R scores are the same as described in the M-SAP. Pre-baseline slope in ALSFRS-R (delta-FRS) is defined as 48 minus the baseline ALSFRS-R total score then divided by the number of months from onset of symptomatic weakness to the Baseline Visit. The number of months will be calculated as the difference in days from onset of symptomatic weakness to the Baseline Visit multiplied by 12 / 365.25. The date of onset of symptomatic weakness will be imputed as the fifteenth day of a month if not specified more precisely.

ALSFRS-R domain scores are exploratory measures of the primary efficacy endpoint ALSFRS-R total score.

#### **5.2** SVC

The derivation of SVC percent-predicted of normal is the same as described in the M-SAP with age calculated as number of days from date of birth to the date of a given SVC assessment divided by 365.25 and with the following correspondence between self-identified race and race defined by Global Lung Initiative (GLI) classification:

| Self-identified Race | GLI-defined Race |
|-------------------------------------------|------------------|
| American Indian or Alaska Native | Mixed/Other |
| Asian | South East Asian |
| Black or African American | African American |
| Native Hawaiian or Other Pacific Islander | Mixed/Other |
| White | Caucasian |
| Unknown | Caucasian |
| Not reported | Caucasian |
| More than one race indicated | Mixed/Other |

### **5.3** Home Spirometry

Home spirometry assesses FVC remotely using a smartphone app (ZEPHYRx, Albany, NY) and a handheld spirometer (Spirobank Smart, Medical International Research, Rome, Italy). Coordinators guide participants through 3 to 8 maneuvers with live-video coaching using the ZEPHYRx platform. Flow loops are classified for acceptability and repeatability using American Thoracic Society (ATS) criteria and are manually reviewed by the NEALS Outcomes Center (Barrow Neurological Institute, Phoenix, AZ). The maximum FVC accepted by the NEALS Outcomes Center is converted to percent of predicted normal using GLI norms based on sex, age at time of assessment, height at time of screening, and race. Age is calculated as number of days from date of birth to the date of a given home spirometry assessment divided by 365.25. Higher values indicate greater respiratory function.

### 5.4 HHD and Grip Strength

The derivation of HHD upper and lower extremity scores and HHD0 are the same as described in the M-SAP with the revision that HHD0 is a composite endpoint with death or death equivalent, whichever occurs first.


A second HHD time-to-event endpoint is defined as the time from the Baseline Visit to the second post-baseline occurrence of a muscle with a strength recording of 0 among those muscles that were non-zero at baseline or time to death or death equivalent, whichever occurs first  $(HHD0^2)$ .

Time at risk for HHD0 and HHD0<sup>2</sup> will be censored at the last date at an HHD assessment was performed up to the end of the Week 24 Visit window.

HHD global average percentage, HHD0, and  $HHD0^2$  are exploratory measures of the secondary endpoint HHD and grip strength.

#### 5.5 Quantitative Voice Characteristics

Voice samples will be collected using the Aural Analytics app installed on either an Android or iOS-based smartphone. At each assessment, participants perform a set of speaking tasks: reading 5 prespecified sentences, reading 5 sentences chosen at random from a large sentence bank, repeating a consonant-vowel sequence, producing a sustained phonation, and counting on a single breath. Speech analysis will be performed by Aural Analytics to derive the following quantitative voice characteristics: maximum phonation time, pause rate, breathy vocal quality, pitch instability, regulation of voicing, articulatory precision, speaking rate, articulation rate, and monotonicity. Aural Analytics will use data on quantitative voice characteristics and participant age, sex, race, height, and weight to derive a prediction of vital capacity at the Baseline Visit.

### 5.6 Biofluid Biomarkers of Neurodegeneration

Blood biomarkers of neurodegeneration, including biomarkers of neuromuscular dysfunction, will be assayed. These will include serum creatinine and serum and CSF neurofilament light chain (NfL). Serum creatinine will be assayed by the kinetic Jaffe method (test 001370, Labcorp, Burlington, NC). NfL will be assayed by single-molecule array (Simoa; Quanterix, Billerica, MA). Levels of serum and CSF NfL that are reported to be below the limit of quantitation will be imputed at the limit of quantitation. Levels of serum and CSF NfL will be log-transformed in all analyses.

#### 5.7 ALSAO-40

The description of the ALSAQ-40 instrument and item-level scores are the same as described in the M-SAP. Each of the five domains will be scored as the mean of all domain-specific items multiplied by 25 (range 0 to 100). An overall symptom index (SI) will be scored as the mean of the five domain scores. A domain score will be missing if more than 20% of the items are missing; otherwise, item non-response will be mean-imputed from other completed items from the same assessment. The ALSAQ-40 SI will be missing if any domain scores are missing. Higher scores indicate worse quality of life.

#### 5.8 CNS-BFS

The definition of CNS-BFS total score is the same as described in the M-SAP.

#### 5.9 Survival

The primary definition of survival time is the same as described in the M-SAP with the clarification that PAV is defined as more than 22 hours per day of noninvasive or invasive

mechanical ventilation for more than seven consecutive days. The date of PAV initiation, where applicable, will be imputed as the fifteenth day of a month if not specified more precisely. A secondary survival endpoint of death alone, independent of any death equivalent, is also defined.

Time at risk for the composite endpoint of death or death equivalent and time at risk for the endpoint of death alone will be measured from each participant's Baseline Visit. Time at risk will be censored at two time points: (1) at the Week 24 Visit as defined in the M-SAP, and (2) at a subsequent assessment of death or death equivalent scheduled approximately at the end of placebo-controlled follow-up of the last RGB participant. The primary analysis of survival will evaluate PAV-free survival to the Week 24 Visit time point.

## 5.10 King's ALS Clinical Staging System

The King's ALS Clinical Staging System (Roche et al. 2012) is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction and levels 4a and 4b indicating nutritional or respiratory failure secondary to ALS, respectively.

Participants will be classified to King's stage 1, 2, 3, 4a, or 4b based on scores from ALSFRS-R assessments according to a published derivation (Balendra et al. 2014). Bulbar involvement is defined as a score less than 4 on any of the ALSFRS-R questions in the bulbar domain (questions 1, 2, and 3). Upper limb involvement is defined as a score less than 4 on either of the ALSFRS-R questions related to hand function (questions 4 and 5A). Lower limb involvement is defined as a score less than 4 on the ALSFRS-R question about walking (question 8). Nutritional failure is defined as responding that the participant uses gastrostomy for greater than 50% of their nutrition. Respiratory failure is defined as a score of 0 on the ALSFRS-R question addressing dyspnea (question 10 or R-1) or a score less than 4 on the ALSFRS-R question about use of mechanical ventilation (question 12 or R-3). Participants without evidence by ALSFRS-R scores of involvement of any of the three central nervous system regions will be scored as King's stage 1 due to their confirmed diagnosis with ALS. Participant may meet criteria for both King's stage 4a and 4b.

### 5.11 Hospitalization and Other Clinical Events

Times to the following clinically relevant events are defined:

- Time to first hospitalization due to a serious adverse event (SAE),
- Time to first hospitalization due to an ALS-related SAE,
- Time to first use of assisted ventilation,
- Time to first placement of a feeding tube,
- Time to King's stage 4a or 4b, and
- Time to first instance of hospitalization for an SAE, feeding tube placement, tracheostomy, initiation of PAV, or death.

Time at risk for each event will be measured from each participant's Baseline Visit. Time to first hospitalization excludes hospitalizations for elective procedures. ALS-related SAEs are those indicated as related to ALS disease progression by the site investigator. Participants who are already using assisted ventilation or have a feeding tube at the time of the Baseline Visit will be

excluded from analysis of those endpoints. Death or death equivalent will be considered an outcome for each of the events listed, forming a composite endpoint.

Time at risk for these events will be censored at the Week 24 Visit, if completed, the date of consent withdrawal, if withdrawn, or the last date at which the status of each endpoint is known prior to the end of the Week 24 Visit window for participants lost to follow-up. Time to King's stage 4a or 4b is interval censored between ALSFRS-R assessments.

### 5.12 Pharmacodynamic Biomarkers

Myeloperoxidase protein and activity levels in plasma samples collected at Baseline and Weeks 4, 8, 16, and 24 will be assayed among participants randomized to active treatment. Details of the assay techniques will be specified when known.

### **5.13 Clinical Safety Laboratory Tests**

Clinical safety labs include hematology, blood chemistry panel, liver function tests, thyroid function, urinalysis, and pregnancy testing in women of childbearing potential as specified in Section 9.1.2 Clinical Safety Laboratory Tests of the Master Protocol:

- Hematology: hematocrit, hemoglobin, platelet count, red blood cell (RBC) count, mean
  corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin
  concentration, RBC distribution width (RDW), RBC morphology, white blood cell (WBC)
  count, and counts and percentages of basophils, eosinophils, lymphocytes, monocytes, and
  neutrophils;
- Blood chemistry panel: bicarbonate, chloride, potassium, sodium, calcium, magnesium, phosphate, blood urea nitrogen, creatinine, estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) four-variable equation, creatinine clearance calculated using the Cockcroft-Gault equation, and glucose;
- Liver function tests: alanine aminotransferase (ALT [SGPT]), aspartate aminotransferase (AST [SGOT]), alkaline phosphatase (ALP), albumin, total protein, total bilirubin (TBL);
- Thyroid function tests: thyroid-stimulating hormone (TSH), reflex T3 and T4 when TSH levels are abnormal;
- Urinalysis: clarity, color, specific gravity, pH, microalbumin, protein, glucose, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase, and blood; and
- Pregnancy: qualitative and quantitative serum human chorionic gonadotropin (hCG).

Clinical safety labs will also include derived measures of potential drug-induced liver injury (DILI), including those that potentially meet the Hy's law criteria, as distinct safety lab outcomes.

Three potential DILI criteria will be defined:

- ALT or AST >3x ULN with TBL >1.5x ULN
- AST or ALT >3x ULN with TBL >2x ULN
- AST or ALT >3x ULN with TBL >2x ULN and ALP <2x ULN (potential Hy's Law cases) where ULN is upper level of normal and all levels are measured on the same day.


### 6. Statistical Methodology

### 6.1 Analysis Sets

The ITT analysis set is henceforth referred to as the Full Analysis Set (FAS) and defined as follows:

• Full Analysis Set (FAS): Participants who were randomized within RGB plus placebo participants from specified regimens, classified according to their randomized treatment assignment. Observations made after premature permanent discontinuation of study drug are included in this sample, should such participants remain on study. Observations completed after regimen data lock are excluded. Participants determined to not meet ALS diagnostic criteria are excluded.

The definition of the STF analysis set is revised as follows:

Safety Full (STF) Set: Participants who initiated treatment within RGB plus placebo
participants from specified regimens who are not known to be ineligible for RGB and who
initiated treatment in their respective regimen, classified according to the treatment they
actually received. Observations made after premature permanent discontinuation of study
drug are included in this sample, should such participants remain on study. Observations
completed after regimen data lock are excluded.

An analysis set restricting shared placebo participants to those regimens in which study drug is administered by the same route as RGB is defined as follows:

• Efficacy Common Mode of Administration (ECM) Set: The subset of participants in the FAS analysis set who are in regimens in which study drug is administered by the same route as RGB.

The definitions of the ECC, ERO, STN, and SRO analysis sets are the same as described in the M-SAP with reference to the ITT analysis set now referencing the FAS analysis set. The following analysis set is specific to RGB:

Efficacy Per-protocol (EPP) Set: The subset of participants in the FAS analysis set who initiated study treatment and who were not involved in protocol deviations that affected the scientific integrity of the trial as documented prior to data lock, classified according to the treatment they actually received. Inclusion or exclusion from the EPP analysis set of any participant for whom treatment assignment was unblinded prior to data lock will be governed by the prespecified criteria above. If a participant's data is truncated for inclusion in the EPP analysis set due to non-adherence to protocol-specified dosing, clinical events observed up to 28 days after the censoring event will be included in the EPP analysis set. For all other events leading to truncation of a participant's data, no events beyond that date will be included. Data from placebo participants shared from other regimens will not be truncated due to non-adherence to protocol-specified dosing.

•

Applicable analysis sets (FAS, ECM, EPP, STF, and STN) will include shared placebo participants from regimens A and C only. Data from shared placebo participants will include visits and events that occurred on or before the date of the final placebo-controlled period follow-up of a regimen A, B, or C participant. As only concurrently enrolling regimens are

contributing to efficacy analyses, the FAS and ECC analysis sets are synonymous and only the FAS analysis set will be referenced. As regimen A is administered by subcutaneous injection and regimen C is administered orally, only regimen C will contribute shared placebo participants for the ECM and STN analysis sets.

### 6.2 Baseline Characterization

The baseline characteristics summarized for participants randomized within RGB are the same as specified in the M-SAP with the addition of ALSAQ-40 domain scores and SI, CNS-BFS total score, King's stage, weight, body mass index (BMI), serum urate concentration, serum creatinine concentration, and serum NfL concentration.

### 6.3 Primary Efficacy Analysis and Supportive Analyses

The primary analysis for RGB is a Bayesian shared-parameter, repeated-measures model of ALSFRS-R that accounts for loss of follow-up due to mortality. Details of the model, including documentation of operating characteristics under a range of scenarios, are provided in the "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (Appendix 1 to the Master Protocol). The Bayesian shared-parameter, repeated-measures model will be applied to the FAS analysis set as the primary analysis, to the ECM and ERO analysis sets as sensitivity analyses, and to the EPP analysis sets as a supportive analysis.

The estimand of the primary analysis is the relative rate of disease progression (the "disease rate ratio" or DRR) of active treatment relative to placebo in the FAS population under an assumption that active treatment slows mean time to death or death equivalent by the same proportion as treatment slows the mean rate of functional progression as measured by change in ALSFRS-R total score over time. The estimand is defined by the following attributes:

- Treatment: verdiperstat administered orally at a dosage of 600 mg BID vs. placebo.
- Population: FAS population as defined in Section 6.1.
- Variables: time to death or death equivalent and rate of change in ALSFRS-R total score from baseline to the Week 24 Visit.
- Intercurrent event 1: treatment discontinuation due to death: no ALSFRS-R data from participants who reach the death or death equivalent endpoint are included in the analysis, handled via mortality component in model, composite variable strategy approach.
- Intercurrent event 2: treatment discontinuation not due to death: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation regardless of concomitant medication, for those participants who have not been censored due to mortality. Missing data post-treatment will not be imputed, handled via missing at random assumption.
- Population-level summary: mean ratio of hazard or progression rate of active treatment relative to placebo.

### 6.4 Interim Analysis

RGB will be considered for early stopping for futility according to the interim analysis schedule and definition specified in the "ALS Master Protocol Recommended Statistical Analysis, Design

and Simulation Report" (Appendix 1 to the Master Protocol). RGB will not be stopped early for success.

## 6.5 Secondary Efficacy Analyses

## 6.5.1 Hierarchical Testing

Primary inference for secondary efficacy endpoints will be based on analysis of the FAS analysis set using a repeated-measures linear mixed model for functional endpoints (see Section 6.5.2 below) and by Kaplan-Meier product-limit estimates and log-rank test for the primary survival endpoint (see Section 6.5.4 below). The sequence for testing secondary efficacy endpoints is the following:

- 1. HHD upper extremity percentage,
- 2. SVC,
- 3. HHD lower extremity percentage, and
- 4. Survival.

If the primary analysis indicates a significant slowing in disease progression from the Bayesian shared-parameter, repeated-measures model of ALSFRS-R and mortality, then each secondary efficacy endpoint in succession would be declared significant in the specified sequence using a comparison-wise criterion of two-tailed p < 0.05. After the first failure to declare significance, no endpoints lower in the hierarchy can be significant. This sequential closed-testing procedure controls the overall type 1 error rate at 5%. Nominal comparison-wise p-values for secondary efficacy endpoints will also be reported.

## 6.5.2 Repeated-measures Model

The specification of the repeated-measures linear mixed model and the primary linear contrast for estimating differences in 24-week change from baseline in a given continuous efficacy endpoint (ALSFRS-R total and domain scores, HHD upper extremity, lower extremity, and global average percentages, SVC, FVC by home spirometry, serum creatinine, serum NfL, ALSAQ-40 domain scores and SI, and CNS-BFS total score) are revised from those specified in the M-SAP to include a main effect of treatment.

The model will include fixed terms for discrete visit, treatment group, treatment group  $\times$  visit interaction, centered time since symptom onset and centered time since symptom onset  $\times$  visit interaction, centered delta-FRS and centered delta-FRS  $\times$  visit interaction, centered baseline riluzole use and centered baseline riluzole  $\times$  visit interaction, and centered baseline edaravone use and centered baseline edaravone  $\times$  visit interaction. The following equations describe the model with regimen random effects:

$$Y_{ij} = a_{k(i)} + \gamma_1 t_i + \gamma_{2,j} v_j + \gamma_3' \mathbf{z}_i + \gamma_{4,j} t_i v_j + \gamma_{5,j}' \mathbf{z}_i v_j + \epsilon_{ij}$$

$$a_k \sim N(0, \sigma_r^2), \, \boldsymbol{\epsilon}_{i \cdot} \sim N(\mathbf{0}, \mathbf{R}), \, \text{Cov}(b_{k(i)}, \epsilon_{ij}) = 0$$
(eqn. 1)

where  $Y_{ij}$  is a given efficacy endpoint measured in participant i at visit j,  $a_{k(i)}$  is a random intercept for regimen k to which participant i was assigned,  $v_j$  is an indicator variable for visit j,  $z_i$  is the vector of covariates (centered time since onset, centered delta-FRS, centered baseline riluzole use, and centered baseline edaravone use) for participant i,  $t_i$  is an indicator variable for treatment t to which participant t was assigned,  $v_i$ ,  $v_i$ ,  $v_j$ ,  $v_j$ ,  $v_j$ , and  $v_i$  are estimated parameters

and vectors of parameters for the fixed effects, and  $\epsilon_{ij}$  is the residual for participant i at visit j. The regimen-specific random effects are normally distributed with mean 0 and variance  $\sigma^2_r$ . The vector of residuals for a given participant are normally distributed with mean 0 and an unstructured covariance matrix  $\mathbf{R}$ . The regimen-specific random effect for a given participant and residuals for that participant are uncorrelated.

The following SAS code specifies the model:

where id is a participant study identifier, trtrnd is the randomly assigned treatment group, visit is the visit identifier, Value is value of the efficacy endpoint being tested for a given participant at a given visit, sx2b1 is years since ALS symptom onset centered at the sample median, dFRS is pre-baseline slope centered at the sample median, r1z is an indicator of riluzole use at baseline, and edv is an indicator of edaravone use at baseline. The primary estimate will be the treatment-dependent difference in change from baseline to the Week 24 Visit. The estimate and its 95% Wald confidence bounds will be obtained by a linear contrast of adjusted means. The following SAS code specifies the linear contrast for a regimen with one active treatment assuming an endpoint measured every 8 weeks and that the sort order for treatment group has the active group last and visits are sorted chronologically:

```
estimate "3|Act vs Plb|dWk 24" trtrnd*visit 1 0 0 -1 -1 0 0 1 / cl;
```

A significant difference in 24-week change from baseline in the direction of greater improvement or less worsening among participants randomized to active treatment would support inference of benefit from active treatment for the efficacy endpoint being tested.

The estimand estimated by the primary linear contrast of the repeated-measures linear mixed model is the mean difference in 24-week change from baseline of a given continuous efficacy endpoint in the active treatment group relative to the placebo group in the FAS population. The estimand is defined by the following attributes:

- Treatment: verdiperstat administered orally at a dosage of 600 mg BID vs. placebo.
- Population: FAS population as defined in Section 6.1.
- Variables: absolute change in endpoint from baseline to the Week 24 Visit.
- Intercurrent event: treatment discontinuation: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation. Missing data post-treatment, including data missing due to death, will not be imputed, handled via missing at random assumption.
- Population-level summary: difference in conditional means of active treatment relative to placebo.

Inference from this analysis is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and is the primary analysis for secondary

endpoints. A separate supportive analysis will include centered baseline serum NfL level and the interaction of centered baseline serum NfL level and visit as additional covariates.

### 6.5.3 Random-slopes Model

The specification of the random-slopes linear mixed model and the primary linear contrast for estimating differences in mean rate of progression in a given continuous efficacy endpoint (ALSFRS-R total and domain scores, HHD upper extremity, lower extremity, and global average percentages, SVC, FVC by home spirometry, quantitative voice characteristics, serum creatinine, serum NfL, ALSAQ-40 domain scores and SI, and CNS-BFS total score) are revised from those specified in the M-SAP to include a main effect of treatment and to specify that study months are calculated as the difference in days from the Baseline Visit to the date of assessment of a given endpoint multiplied by 12 / 365.25.

The model will include fixed terms for month since the Baseline Visit, treatment group, treatment group × month interaction, centered years since ALS symptom onset and centered years since ALS symptom onset × month interaction, centered delta-FRS and centered delta-FRS × month interaction, centered baseline riluzole use and centered baseline riluzole use × month interaction, and centered baseline edaravone use and centered baseline edaravone use × month interaction. The following equations describe the model with regimen random effects:

$$Y_{ij} = \gamma_1 + a_{k(i)}^0 + b_i^0 + \gamma_2 t_i + \gamma_3' \mathbf{z}_i$$

$$+ \left(\gamma_4 + a_{k(i)}^1 + b_i^1 + \gamma_5 t_i + \gamma_6' \mathbf{z}_i\right) m_{ij} + \epsilon_{ij}$$

$$\{a_k^0, a_k^1\} \sim N(\mathbf{0}, \mathbf{\Sigma}_r), \{b_k^0, b_k^1\} \sim N(\mathbf{0}, \mathbf{\Sigma}_p), \epsilon_{ij} \sim N(\mathbf{0}, \sigma_\epsilon^2)$$

$$Cov(\mathbf{a}_k, \mathbf{b}_k) = \mathbf{0}, Cov(\mathbf{a}_k, \boldsymbol{\epsilon}_{i\cdot}) = \mathbf{0}, and Cov(\mathbf{b}_k, \boldsymbol{\epsilon}_{i\cdot}) = \mathbf{0}$$
(eqn. 2)

where  $Y_{ij}$  is a given efficacy endpoint measured in participant i at visit j,  $a^0_{k(i)}$  and  $a^1_{k(i)}$  are random intercept and slope for regimen k to which participant i was assigned,  $b^0_i$  and  $b^1_i$  are random intercept and slope for participant i,  $z_i$  is the vector of covariates (centered time since onset, centered delta-FRS, centered baseline riluzole use, and centered baseline edaravone use) for participant i,  $m_{ij}$  is the time from baseline to observation j for participant i in months calculated as days x 12 / 365.25,  $t_i$  is an indicator variable for treatment t to which participant i was assigned,  $\gamma_1$ ,  $\gamma_2$ ,  $\gamma_3$ ,  $\gamma_4$ ,  $\gamma_5$ , and  $\gamma_6$  are estimated parameters and vectors of parameters for the fixed effects, and  $\epsilon_{ij}$  is the residual for observation j for participant i. The regimen-specific random effects are normally distributed with mean  $\mathbf{0}$  and unstructured covariance matrix  $\mathbf{\Sigma}_r$ . The participant-specific random effects are normally distributed with mean  $\mathbf{0}$  and unstructured covariance matrix  $\mathbf{\Sigma}_p$ . The residuals for a given participant are normally distributed with mean  $\mathbf{0}$  and variance  $\sigma^2_{\epsilon}$ . The regimen-specific random effects, participant-specific random effects, and residuals are uncorrelated.

The following SAS code specifies the model:

where month is time in months from the Baseline Visit (assuming 12 months in an average of 365.25 days per year) and other fields are the same as identified above in Section 6.5.2. The primary estimand will be the treatment-dependent difference in slopes. The estimate and its 95% Wald confidence bounds will be obtained by a linear contrast of adjusted means. The following SAS code specifies the linear contrast for a regimen with one active treatment assuming that the sort order for treatment group has the active group last:

```
estimate "3|Act vs Plb|Slope (/mn)" month 0 trtrnd*month -1 1 / cl;
```

A significant difference in slopes in the direction of greater improvement or less worsening among participants randomized to active treatment would support inference of benefit from active treatment for the efficacy endpoint being tested.

The estimand estimated by the primary linear contrast of the random-slopes linear mixed model is the difference in mean rate of progression of a given continuous efficacy endpoint in the active treatment group relative to the placebo group in the FAS population. The estimand is defined by the following attributes:

Treatment: verdiperstat administered orally at a dosage of 600 mg BID vs. placebo.

Population: FAS population as defined in Section 6.1.

Variables: mean rate of change in endpoint from baseline to the Week 24 Visit.

Intercurrent event: treatment discontinuation: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation. Missing data post-treatment will not be imputed, handled via missing at random assumption.

Population-level summary: difference in conditional mean slopes of active treatment relative to placebo.

Inference from these analyses is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and inference from the repeated-measures linear mixed model for secondary endpoints. A separate supportive analysis will include centered baseline serum NfL level and the interaction of centered baseline serum NfL level and study month as additional covariates.

### 6.5.4 Survival and Time to Clinical Events

Survival and time to hospitalizations and clinical events will be analyzed in the FAS, ECM, ERO, EPP, STF, SFN, and SRO analysis sets. Survival analyses that include follow-up beyond the placebo-controlled period will be analyzed in the ERO analysis set. The summaries and analyses of time to death or death equivalent are the same as specified in the M-SAP with the revision to include baseline age as an additional covariate in adjusted models, with the addition that the endpoints of time to death independent of occurrence of death equivalents and time to each of the hospitalization and clinical events will be separately analyzed using the same models, and with an additional adjusted analysis that includes baseline serum NfL level as a covariate. Analysis of time to King's stage 4a or 4b will accommodate interval censoring between ALSFRS-R assessments and will be stratified by baseline King's stage.

#### 6.5.5 CAFS

The primary CAFS analysis is as specified in the MPRDR. Additional, unadjusted CAFS analyses are the same as specified in the M-SAP, including specification that pair-wise comparison of change in ALSFRS-R total score for participants who cannot be ranked by time to death or death equivalent is to the maximum follow-up time at which both participants have an observation, and with the following additions:

- 1. HHD upper and lower extremity percentage and SVC will be analyzed by CAFS by substituting change from baseline for those secondary efficacy endpoints in place of ALSFRS-R total score,
- 2. An additional set of CAFS analyses will use multiple imputation to extend follow-up of ALSFRS-R total score, HHD upper and lower extremity percentage and SVC for participants who early terminate, withdraw consent, or are lost to follow-up,
- 3. An additional set of CAFS analyses for ALSFRS-R total score, HHD upper and lower extremity percentage and SVC will use time to death alone independent of any death equivalent,
- 4. An additional set of CAFS analyses for ALSFRS-R total score, HHD upper and lower extremity percentage, and SVC will adjust rank scores in a linear model with the following covariates: time from ALS symptom onset, delta-FRS, baseline use of riluzole, and baseline use of edaravone, and
- 5. An additional set of CAFS analyses for ALSFRS-R total score, HHD upper and lower extremity percentage, and SVC will adjust rank scores in a linear model with the following covariates: time from ALS symptom onset, delta-FRS, baseline use of riluzole, baseline use of edaravone, and baseline serum NfL level.

The multiple imputation model used to extend follow-up of functional scores for participants who early terminate, withdraw consent, or are lost to follow-up will use linear regression with covariates of time since symptom onset, delta-FRS, baseline riluzole use, baseline edaravone use, and each observed functional score prior to a missing assessment.

Inference from CAFS analyses is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary outcome and supportive of inference from the repeated-measures model for the secondary outcomes of HHD upper extremity score, SVC, and HHD lower extremity score. Primary inference from CAFS analyses will compare survival by time to death or death equivalent, will compare change in function to the last jointly observed time point, and will adjust for the specified covariates.

#### **6.5.6** HHD0 and HHD0<sup>2</sup>

Analyses of HHD0 are the same as specified in the M-SAP with the addition of parallel analyses of HHD0<sup>2</sup>, with a separate analysis that includes baseline serum NfL level as an additional covariate, and with the clarification that time to zero strength for both analyses is interval censored between HHD assessments.

Inference from these analyses is supportive of inference from the repeated-measures linear mixed model for HHD upper and lower extremity scores.

#### **6.5.7** Quantitative Voice Measures

Given the high frequency of voice recordings, a repeated-measures analysis with unstructured covariance is overly flexible but the assumption of linear change required by the random-slopes

model may be overly rigid. To complement estimates from the random-slopes linear mixed model, quantitative voice characteristics will be analyzed in a linear mixed model in which the temporal profile for both fixed and random terms is modeled using cubic B-splines with knots at 8 and 16 weeks. The model will include fixed terms for B-splines (4 terms), treatment group (2 levels), treatment group × B-spline interaction, centered time since symptom onset and centered time since symptom onset × B-spline interaction, centered delta-FRS and centered delta-FRS × B-spline interaction, centered baseline riluzole use and centered baseline riluzole × B-spline interaction, and centered baseline edaravone use and centered baseline edaravone × B-spline interaction The model will include random regimen-specific intercepts and slopes with unstructured covariance, random participant-specific B-splines (5 terms) with unstructured covariance, and a first-order autoregressive structure for residuals. A simplified covariance structure assuming no regimen-level covariance, heterogeneous compound symmetric covariance among the random B-splines, conditional independence of residuals, or a combination of the three simplifying assumptions will be used if the full model fails to converge. The primary estimand will be the treatment-dependent difference in 24-week change from baseline. The estimate and its 95% Wald confidence bounds will be obtained by a linear contrast of adjusted means. A separate analysis will include centered baseline serum NfL level and the interaction of centered baseline serum NfL level and B-splines as additional covariates.

### 6.5.8 Placebo Multiple Imputation

Placebo multiple imputation analyses are the same as specified in the M-SAP and will be applied to ALSFRS-R total score, HHD upper and lower extremity percentages, and SVC.

The following SAS code specifies the imputation for an endpoint measured every 8 weeks:

where Wk00, Wk08, Wk16, and Wk24 are the values of a given efficacy endpoint at the Baseline, Week 8, Week 16, and Week 24 Visits, respectively, trtnd has a value of zero (0) for participants randomized to placebo, and x and y take appropriate values to specify the range of a given outcome measure (i.e., 0 and 48 for ALSFRS-R total score; 0 and . for HHD upper and lower extremity percentages and SVC).

Inference from these analyses is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and assess sensitivity to the missing data assumption of the repeated-measures linear mixed model for secondary endpoints in the FAS analysis set. A separate analysis will include centered baseline serum NfL level as an additional covariate in both imputation stages.

### 6.5.9 Additional Sensitivity Analyses of Primary and Key Secondary Outcomes

Sensitivity analyses of primary and key secondary efficacy outcomes are the same as specified in the M-SAP.

### 6.5.10 Subgroup Analyses

In addition to the subgroups specified in the M-SAP, the following additional subgroups will be analyzed in the random-slope model (see Section 6.5.3) for primary and secondary efficacy endpoints in the FAS analysis set:

- Baseline use of riluzole and edaravone (neither, riluzole only, edaravone only, both),
- Age (less than 65 years vs. 65 years or older),
- Sex (female vs. male),
- Race (white vs. any minority race with greater than 5% prevalence in the sample),
- Ethnicity (Hispanic or Latino vs. non-Hispanic or Latino),
- Weight (less than 70 kg, 70 to less than 85 kg, 85 kg or more),
- BMI (less than  $18.5 \text{ kg/m}^2$ ,  $18.5 \text{ to less than } 25 \text{ kg/m}^2$ ,  $25 \text{ kg/m}^2$  or more),
- Chronic kidney disease (CKD) stage (stage 1 or better [eGFR 90 mL/min/1.73m<sup>2</sup> or more], stage 2 [eGFR 60 to 89 mL/min/1.73m<sup>2</sup>], stage 3 or worse [eGFR less than 60 mL/min/1.73m<sup>2</sup>]),
- Time since onset of weakness (less than 18 months vs. 18 months or longer),
- Baseline serum NfL concentration (by median split), and
- Site (individual sites with at least 5 participants per treatment group and all participants from sites with fewer than 5 participants per treatment group pooled).

For each classification, unknown, not reported, and missing will be considered one group. All individuals not included in a specified subgroup will be combined into a mixed, "other" group. The "other" group will be included in analyses if its prevalence is greater than 5%; otherwise, the "other" group will be excluded.

In cases where a model for a given subgroup and endpoint fails to converge, the covariance terms for the regimen-specific random effects will be simplified from unstructured covariance of intercepts and slopes to separate, uncorrelated variance components for intercepts and slopes. If convergence still fails, regimen-specific intercepts and slopes will be modeled as fixed effects. If convergence still fails, the participant-specific random effects will be simplified from unstructured covariance of intercepts and slopes to separate, uncorrelated variance components for intercepts and slopes.

### 6.5.11 Comparison of Controls across Regimens

Comparisons of placebo participants across regimens are the same as specified in the M-SAP with separate analyses that include baseline serum NfL level as an additional covariate in adjusted analyses plus applicable interaction terms as relevant to a given model.

#### **6.5.12 Pharmacokinetic Analyses**

Pre-dose concentrations of verdiperstat in plasma will be summarized by treatment group and visit in the ERO sample. Concentrations below the limit of quantitation (BLQ) will be replaced with one half of the lower limit of quantitation. Summaries will include number of observations, number and percentage with concentrations BLQ, arithmetic mean, median, standard deviation, minimum, maximum, geometric mean, geometric coefficient of variation (calculated as sqrt(exp(variance of log-transformed concentrations) – 1)), and 95% confidence bounds for the geometric mean assuming log-normally distributed data.

Plasma concentration data of verdiperstat may be subjected to population pharmacokinetic analysis to derive population estimates of pharmacokinetic parameters and test the effect of various covariates such as age, weight, and sex. Details of the analysis will be described in a separate data analysis plan (DAP). This analysis may be performed by combining data from the current study with data from other studies of verdiperstat, if deemed appropriate. The population pharmacokinetic analysis will be performed by Biohaven and reported in a separate modelling report.

### 6.5.13 Pharmacodynamic Biomarker Analyses

Change in myeloperoxidase protein and activity levels in plasma will be summarized by treatment group and visit in the ERO sample. Summary statistics will be provided for the values, change from baseline, and percent change from baseline at each scheduled assessment time point. Myeloperoxidase protein and activity levels in plasma will be analyzed in a repeated-measures linear mixed model that includes fixed terms for visit, time from last dose of verdiperstat, and time from last meal.

## 6.6 Safety Analyses

#### **6.6.1** Treatment-emergent Adverse Events

Summaries and analyses of treatment-emergent adverse events (TEAE) are the same as specified in the M-SAP with the following revisions.

TEAEs are defined as those adverse events with onset dates in the interval from double-blind treatment initiation to the earliest of the Final Safety Visit, the date the participant dies, early terminates, or is lost to follow-up, 28 days after last dose of study drug, or the date of first dose of study drug during participation in the OLE, if so exposed. Adverse events with onset on the day of double-blind treatment initiation and adverse events with incompletely specified onset date where the ambiguous date spans the day of double-blind treatment initiation or the earliest of the events above that define the end of the treatment-emergence interval will be assumed to be treatment emergent except for those known to precede first exposure to study drug.

In addition to summaries specified in the M-SAP, the following categories of adverse events will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term: (a) all adverse events, including those not classified as TEAEs, (b) fatal TEAEs, and (c) TEAEs that occurred during a participant's COVID-19 infection (defined as 5 days prior to symptom onset to end of COVID-19 symptoms or end of double-blind follow-up, if ongoing).

TEAEs indicating COVID-19 infection are the following: Asymptomatic COVID-19, COVID-19, COVID-19 pneumonia, COVID-19 treatment, Post-acute COVID-19 syndrome, SARS-CoV-

2 antibody test positive, SARS-CoV-2 RNA increased, SARS-CoV-2 sepsis, SARS-CoV-2 test false negative, SARS-CoV-2 test positive, SARS-CoV-2 viraemia, Suspected COVID-19.

Treatment-dependent differences in the proportion of participants experiencing a given type of TEAE will not be tested. Treatment-dependent differences in TEAE incidence rates in units of number per 100 participant years will be estimated as differences rather than ratios, will include comparison-wise 95% confidence intervals with variance estimates obtained by the delta method, and will be provided for overall classes of TEAEs not further classified by MedDRA term (all TEAEs, serious TEAEs, severe TEAEs, TEAEs leading to discontinuation of study drug, TEAEs resulting in death, and TEAEs of special interest) and TEAEs with at least 5% prevalence in the active arm.

Listings will document all adverse events (including those not classified as treatment emergent), TEAEs, serious TEAEs, severe TEAEs, related TEAEs, TEAEs leading to discontinuation of study drug, TEAEs resulting in death, and TEAEs of special interest.

### 6.6.2 Safety Labs

Summaries and analyses of clinical safety labs are the same as specified in the M-SAP with the revision that lab results collected more than 28 days after last dose of study drug will not be tabulated, that abnormal levels will be classified to a toxicity grade based on quantitative grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, and with the addition that maximum toxicity over all post-baseline visits that occur within 28 days or fewer after last dose of study drug will be included in shift tables along with visit-specific shifts.

The proportion of participants with TSH ≥10 mIU/L and the proportion with signs or symptoms of hypothyroidism will be presented as shift tables vs. the status of each participant at baseline for each visit and over all post-baseline visits that occur within 28 days or fewer after last dose of study drug by treatment group in all safety samples. The absolute level and the absolute change from baseline for free T3, free T4, and TSH will be summarized as means, standard deviations, medians, and ranges at each visit by treatment group in all safety samples.

#### 6.6.3 ECG Results

Summaries of ECG parameters and findings are the same as specified in the M-SAP with the revision that ECG parameters and findings collected more than 28 days after last dose of study drug will not be tabulated.

### 6.6.4 Vital Signs and Weight

Summaries and analyses of vital signs and weight are the same as specified in the M-SAP with the revision that vital signs and weight collected more than 28 days after last dose of study drug will not be tabulated.

#### 6.6.5 Suicidality

Summaries of suicidality are the same as specified in the M-SAP with the revision that suicidality noted more than 28 days after last dose of study drug will not be tabulated.

### 6.7 Other Analyses

### 6.7.1 Participant Disposition

All participants consented to the Master Protocol between the time of the first and last consent of a participant assigned to a regimen included in the FAS analysis set will be summarized as a single set for the following events: consented to the Master Protocol, failed screening for the Master Protocol, other reasons not assigned to a regimen (including timing out of the screening window, death, withdrawal of consent, early termination, and administrative termination), and assigned to a regimen. Reasons for Master Protocol screen failure will be summarized.

All participants in the above sample assigned to a regimen will be summarized as two sets (final screening for RGB vs. final screening for a non-RGB regimen) for the following events: consented to a regimen, failed screening for a regimen, other reasons not randomized within a regimen (including timing out of the screening window, death, withdrawal of consent, early termination, and administrative termination), and randomized within a regimen. If a given individual is screened multiple times prior to randomization within a regimen, then the final screening experience of that individual will be summarized. Reasons for RGB screen failure will be summarized separately for all participants screened for RGB whether that was their final screening experience or not.

All participants in the FAS analysis set will be summarized as two sets (randomization to active study drug vs. randomization to placebo) for the following events: initiated regimen-specific study drug, prematurely terminated study participation due to death, withdrawal of consent, early termination, loss to follow-up, or administrative termination, completed 24-week follow up, and completed a safety follow-up visit vs. continued into the OLE. Reasons for withdrawal of consent or early termination after randomization will be summarized.

Any randomized participants excluded from the FAS and EPP analysis sets or included in the FAS analysis set but not contributing to the primary analysis will be identified in a listing together with the reason for their exclusion.

### 6.7.2 Study Drug Compliance and Tolerance

Summaries of study drug compliance and tolerance are the same as specified in the M-SAP with the clarification that summaries will be reported for the ERO and SRO analysis sets and that date of permanent discontinuation of study drug is the date of last use of double-blind study drug among all participants in a given analysis set.

The number of days of exposure to study drug will be calculated in three ways:

- as the number of days from dose initiation to the final safety assessment during the placebocontrolled period, inclusive,
- as the number of days from dose initiation to drug withdrawal, inclusive, less any interval during which use of study drug was interrupted (individual missed doses will not be subtracted unless noted in the dosage management log), and
- as the number of days from dose initiation to the earlier of final contact during the placebocontrolled period or 28 days after last dose of study drug, inclusive.


The proportion of participants who interrupted study drug or reduced study drug dosage and the time to first study drug interruption or dosage reduction will be summarized. The number of days of exposure to a reduced dosage of study drug will be summarized.

#### **6.7.3** Concomitant Medication Use

Summaries of concomitant medication use are the same as specified in the M-SAP with the clarification that medications taken at baseline and those initiated after first dose of study drug will be separately summarized and will be classified by ATC Therapeutic class and WHODrug Preferred base name.

## **6.7.4** Medical History

Medical histories will be summarized by MedDRA system organ class, high level term, and preferred term in the STF and SRO analysis sets.

#### 6.7.5 Blindedness

The proportions of participants and site investigators who report on the Exit Questionnaire a guess of active vs. placebo treatment assignment, each level of surety of that guess, and each of five pre-specified reasons for making a treatment assignment will be summarized by treatment group in the FAS and ERO analysis sets. Treatment-dependent differences in the proportion guessing active treatment assignment will be tested among all respondents and among those stating they are at least somewhat sure of their guess by Fisher's exact test and the difference in proportion guessing active treatment assignment will be estimated with confidence bounds.

#### 6.7.6 Protocol Deviations

The number of major and minor protocol deviations will be summarized by type of deviation and treatment group in all analysis sets. Listings of all protocol deviations will be produced.

### 6.7.7 Impact of COVID-19 Pandemic

The proportions of planned assessments missed due to COVID-19 restrictions or disruptions will be summarized by treatment group, visit, and type of assessment in the FAS and ERO analysis sets. Protocol deviations that resulted from COVID-19 restrictions or disruptions will be summarized by treatment group and type of deviation in the FAS and ERO analysis sets.

A listing will document participants with assessments missed due to COVID-19 restrictions or disruptions and those experiencing protocol deviations that resulted from COVID-19 restrictions or disruptions and will describe the manner affected by COVID-19.

### 7. Validation

#### 7.1 Primary Efficacy Analysis

Validation of the primary efficacy analysis is the same as specified in the M-SAP.

### 7.2 Secondary, Exploratory, and Safety Analyses

Validation of secondary, exploratory, and safety analyses are the same as specified in the M-SAP.

### 8. References

The following references are cited in addition to those specified in the M-SAP:

Balendra R, Jones A, Jivraj N, Knights C, Ellis CM, Burman R, Turner MR, Leigh PN, Shaw CE, Al-Chalabi A. Estimating clinical stage of amyotrophic lateral sclerosis from the ALS Functional Rating Scale. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Jun;15(3-4):279-84.

Roche JC, Rojas-Garcia R, Scott KM, Scotton W, Ellis CE, Burman R, Wijesekera L, Turner MR, Leigh PN, Shaw CE, Al-Chalabi A. A proposed staging system for amyotrophic lateral sclerosis. Brain. 2012 Mar;135(Pt 3):847-52.


# **DocuSign**

#### **Certificate Of Completion**

Envelope Id: 43CE3BBBEB4F402E8E21AC8BC6E110E2

Subject: Please DocuSign: HEALEY ALS Platform RGB R-SAP v3.0 20220722\_unsigned.pdf

Source Envelope:

Document Pages: 34 Certificate Pages: 6

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator: Marianne Chase

mchase@mgh.harvard.edu IP Address: 73.60.69.9

Sent: 7/22/2022 5:56:02 PM

Viewed: 7/22/2022 6:27:23 PM

Signed: 7/22/2022 6:28:00 PM

Sent: 7/22/2022 5:56:03 PM

Resent: 7/24/2022 1:29:19 PM

Resent: 7/24/2022 1:29:34 PM

Resent: 7/24/2022 1:34:02 PM

Viewed: 7/24/2022 2:13:14 PM

Signed: 7/24/2022 2:25:13 PM

### **Record Tracking**

Status: Original

7/22/2022 5:52:11 PM

Holder: Marianne Chase

mchase@mgh.harvard.edu

Location: DocuSign

**Timestamp** 

### **Signer Events**

Ben Saville

ben@berryconsultants.net

Ben Saville

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

**Signature** 

Ben Saville

Signatures: 5

Initials: 0

50221BD2-F3C9-432B-9863-2C6FEC7283AD

Using IP Address: 72.182.14.11

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

### Electronic Record and Signature Disclosure:

Accepted: 6/24/2020 5:24:44 PM

ID: 0826203a-7d83-4395-a4f0-c1a7f44f1ee4

Daniel Campbell

daniel.campbell@biohavenpharma.com

Security Level: Email, Account Authentication

(Required)

Daniel Campbell

Signature Adoption: Pre-selected Style

Signature ID:

C81EA4CB-FB71-4B56-BA19-2BFDD76701C8

Using IP Address: 73.218.27.74

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 3/18/2022 2:26:09 PM

ID: de3203d4-50c7-4436-93af-80d10d5e624b

**Signer Events Signature Timestamp** Eric A. Macklin Sent: 7/22/2022 5:56:02 PM Eric A. Macklin emacklin@mgh.harvard.edu Viewed: 7/22/2022 5:59:57 PM Instructor in Medicine Signed: 7/22/2022 6:00:33 PM Eric Macklin Signature Adoption: Pre-selected Style Security Level: Email, Account Authentication Signature ID: (Required) 8E847DD4-0E85-42A1-B334-DFC089673751 Using IP Address: 173.48.212.201 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 5/8/2020 9:17:52 AM ID: 2308ba7c-abcd-4949-872e-021ea95dc489 Sent: 7/22/2022 5:56:02 PM Merit Cudkowicz Merit (udkowicz cudkowicz.merit@mgh.harvard.edu Viewed: 7/22/2022 7:21:48 PM Chief of Neurology Signed: 7/22/2022 7:22:06 PM Security Level: Email, Account Authentication Signature Adoption: Pre-selected Style (Required), Logged in Signature ID: 9F8FE418-0E50-4C6A-B0A6-7B835E80C644 Using IP Address: 108.26.176.128 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 7/22/2022 7:21:48 PM ID: 607c07a3-ad0a-449c-bd8f-fc576210ec5d -DocuSigned by Sabrina Paganoni Sabrina Paganoni Sent: 7/22/2022 5:56:03 PM Viewed: 7/22/2022 8:37:32 PM Spaganoni@mgh.harvard.edu I approve this document Sabrina Paganoni 07/22/2022 | 5:37:50 PM PDT Signed: 7/22/2022 8:37:53 PM MD PhD MGH 58705BF61CB842A887521BEB826294FA Security Level: Email, Account Authentication (Required), Logged in Signature Adoption: Pre-selected Style Signature ID: 58705BF6-1CB8-42A8-8752-1BEB826294FA Using IP Address: 73.182.245.163 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 7/22/2022 8:37:32 PM ID: 7a43fb4f-8356-4448-ba45-401776d82050 In Person Signer Events Signature **Timestamp Editor Delivery Events Status Timestamp Agent Delivery Events Status Timestamp** 

**Timestamp** 

**Timestamp** 

**Intermediary Delivery Events** 

**Certified Delivery Events** 

**Status** 

**Status** 

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 7/22/2022 5:56:03 PM |
| Certified Delivered | Security Checked | 7/22/2022 8:37:32 PM |
| Signing Complete | Security Checked | 7/22/2022 8:37:53 PM |
| Completed | Security Checked | 7/24/2022 2:25:13 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Insight OBO The Massachusetts General Hospital (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

## Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us

### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### How to contact Insight OBO The Massachusetts General Hospital:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: jhenrique@mgh.harvard.edu

### To advise Insight OBO The Massachusetts General Hospital of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at jhenrique@mgh.harvard.edu and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from Insight OBO The Massachusetts General Hospital

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to jhenrique@mgh.harvard.edu and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

## To withdraw your consent with Insight OBO The Massachusetts General Hospital

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to jhenrique@mgh.harvard.edu and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Insight OBO The Massachusetts General Hospital as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Insight OBO The Massachusetts General Hospital during the course of your relationship with Insight OBO The Massachusetts General Hospital.